CLINICAL TRIAL: NCT07143227
Title: A Randomized, Double-blind, Placebo-controlled Phase Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Dosing of XW003 Injection in Chinese Adolescents With Obesity
Brief Title: A Study of XW003 Injection in Chinese Adolescents With Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCW0502-1111
Record Dates: First submitted 2025-08-13; First posted 2025-08-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-08

CONDITIONS: Obese Adolescents; Obesity
Keywords: Weight management; obesity; XW003; ecnoglutide; glucagon-like peptide-1 (GLP-1); adolescent
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- XW003 Dose 1 (Experimental): once weekly
  Interventions: Drug: XW003 injection
- XW003 Dose 2 (Experimental): once weekly
  Interventions: Drug: XW003 injection
- XW003 Dose 3 (Experimental): once weekly
  Interventions: Drug: XW003 injection
- placebo (Placebo Comparator): once weekly
  Interventions: Drug: placebo with matching volume

INTERVENTIONS:
Drug: XW003 injection — Subcutaneous injection
  Arms: XW003 Dose 1; XW003 Dose 2; XW003 Dose 3
Drug: placebo with matching volume — Subcutaneous injection
  Arms: placebo

SUMMARY:
The aim of the study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of XW003 injection in Chinese adolescents with obesity

DETAILED DESCRIPTION:
In this study, eligible participants will be randomized into one of the three cohorts in a 3:1 ratio to receive either once-weekly subcutaneous XW003 injection or placebo, for up to 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of screening, BMI meets the obesity criteria specified in WS/T586-2018 'screening for overweight and obesity among school-aged children and adolescents', and weight ≥55 kg;
2. At the time of screening, the decrease of body mass index less than 5% after diet and exercise control alone for at least 12 weeks (as reported by participants or parents or legal guardians);

Exclusion Criteria:

1. Pre-adolescent participants (Tanner phase I);
2. Obesity caused by secondary diseases or medications, including: elevated cortisol hormone (e.g. Cushing's syndrome), damage to the pituitary gland and hypothalamus, reduced dosage/discontinuation of weight-loss drugs or monogenic obesity, etc.;
3. Have used any weight-loss drugs, hypoglycemic drugs, or drugs that may cause significant weight gain within 3 months prior to screening;
4. Diagnosis with any type of diabetes;
5. History of acute or chronic pancreatitis, history of gallbladder disease or pancreatic injury

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and severity of adverse events | week 20

SECONDARY OUTCOMES:
Plasma concentrations of XW003 | week 20
Change of body weight from baseline | week 20

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Dr, Principal Investigator — Qilu Hospital of Shandong University; Xinguo Hou, Dr, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No